CLINICAL TRIAL: NCT00927511
Title: A Phase II Study, Comparing a Dose-Titration Regimen of Fulvestrant With the Approved Dosing Regimen in Postmenopausal Patients With Hormone-Responsive Advanced Breast Cancer (ABC) (Fulvestrant Intensity Density Study - Studio FIDeS)
Brief Title: A Study, Comparing a Dose-Titration Regimen of Fulvestrant With the Approved Dosing Regimen in Postmenopausal Patients With Hormone-Responsive Advanced Breast Cancer (ABC)
Acronym: FIDeS
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Regina Elena Cancer Institute (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Paola Papaldo, Regina Elena Cancer Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FIDeS
Record Dates: First submitted 2009-06-24; First posted 2009-06-25 (Estimated); Last update posted 2011-07-22 (Estimated); Status verified 2009-06

CONDITIONS: Breast Cancer
Keywords: metastatic hormone-responsive breast cancer menopausal women
MeSH Terms: conditions — Breast Neoplasms | interventions — Fulvestrant

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- A - Dose Tritation (Experimental): Fulvestrant 500 mg days 0, 14, 28, then 250 mg every 2 weeks for 5 administrations, then 250 mg every 28 days, until progression or unacceptable toxicity
  Interventions: Drug: Fulvestrant
- B- Control (Active Comparator): Fulvestrant 250 mg every 28 days until progression or unacceptable toxicity
  Interventions: Drug: Fulvestrant

INTERVENTIONS:
Drug: Fulvestrant — Fulvestrant 500 mg days 0, 14, 28, then 250 mg every 2 weeks for 5 administrations, then 250 mg every 28 days, until progression or unacceptable toxicity vs Fulvestrant 250 mg every 28 days until progression or unacceptable toxicity
  Other Names: Faslodex

SUMMARY:
In post-menopausal metastatic hormone-responsive breast cancer women.

This study is a two arm randomized trial to evaluate the effectiveness of dose-titration regimen of fulvestrant compared with the approved dosing regimen. Patients will be randomized to one of the following treatment arms:

Arm A: Fulvestrant 500 mg days 0, 14, 28, then 250 mg every 2 weeks for 5 administrations, then 250 mg every 28 days, until progression or unacceptable toxicity Arm B: Fulvestrant 250 mg every 28 days until progression or unacceptable toxicity

DETAILED DESCRIPTION:
Arm A: Fulvestrant 500 mg days 0, 14, 28, then 250 mg every 2 weeks for 5 administrations, then 250 mg every 28 days, until progression or unacceptable toxicity Arm B: Fulvestrant 250 mg every 28 days until progression or unacceptable toxicity

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* Histological or cytological diagnosis of hormone-responsive metastatic breast cancer
* Documented positive hormone receptor status (ER+ve and/or PgR+ve) of primary or metastatic tumor issue, according to the local laboratory parameters
* Postmenopausal women, defined as a woman fulfilling any 1 of the following criteria:
* Age ≥ 60 years
* Age ≥ 45 years with amenorrhoea ≥ 12 months with an intact uterus
* Having undergone a bilateral oophorectomy
* FSH and oestradiol levels in postmenopausal range (utilizing ranges from the local laboratory facility)*

  *In patients who have previously been treated with a monthly LH-RH analogue, the last depot must have been administered more than 13 months (or 15 months in case of 3-monthly LH-RH analogue) prior to randomization, and menses must not have restarted
* Prior hormonal treatment in adjuvant setting is allowed
* No more than one prior hormonal treatment for metastatic disease
* Patients with HER2 positive disease in treatment with specific anti-HER2 therapy (trastuzumab, lapatinib) are allowed
* ECOG performance status 0-2
* Patients fulfilling one of the following criteria:
* Patients with measurable disease as per RECIST criteria. This is defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded) as ≥ 20 mm with conventional techniques or as ≥ 10 mm with spiral CT scan
* Patients with bone lesions, lytic or mixed (lytic + sclerotic), in the absence of measurable disease as defined by RECIST criteria. Bone lesions must be evaluable by plain X-ray, CT or MRI. Patients with lesions identified only on radionucleotide bone scan are not eligible
* Patients with a history of other malignancies are eligible if they have been disease-free for at least 5 years and are deemed by the investigator to be at low risk for recurrence. Patients with the following cancers are eligible if diagnosed and treated within the past 5 years: cervical carcinoma in situ, melanoma in situ, and basal cell or squamous cell carcinoma of the skin
* Patients must have normal organ function as defined below:
* total bilirubin within normal institutional limits
* AST (SGOT)/ALT(SGPT) 2.5 X institutional upper limit of normal
* creatinine within normal institutional limits or creatinine clearance 0.60 mL/min/1.73 m2 for patients with creatinine levels above institutional normal

Exclusion Criteria:

* Receive concurrent treatment with an investigational agent or participate in another clinical trial
* Have a concurrent disease or condition that would make the patient inappropriate for study participation, or any serious medical disorder that would interfere with the patient safety
* Patients with responsive or stable disease after chemotherapy (fulvestrant administration in not allowed as maintenance therapy)
* More than 1 line of chemotherapy in metastatic setting; more than 1 maintenance hormonal therapy
* Life expectancy < 6 months
* Have an active or uncontrolled infection
* Have dementia, altered mental status, or any psychiatric condition that would prohibit the understanding or rendering of informed consent
* History of bleeding diathesis, or long term anticoagulant therapy (other than antiplatelet therapy and low dose warfarin)
* History of hypersensitivity to active or inactive excipients of Fulvestrant

Ages: 45 Years to 85 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Estimated)
Dates: Start 2008-10; Primary Completion 2012-04 (Estimated); Study Completion 2012-04 (Estimated)

PRIMARY OUTCOMES:
Time to progression (sec. RECIST) or death from any cause; where there is no evidence of progression, TTP will be right-censored at last patients contact where status was recorded | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Paola Papaldo, MD, Principal Investigator — Regina Elena Cancer Institute
Locations (1):
- Regina Elena Cancer Institute, Rome, RM, Italy